CLINICAL TRIAL: NCT04325698
Title: A RANDOMIZED, DOUBLE-BLIND BRIDGING SAFETY AND EFFICACY STUDY OF PF-06439535 (CN) PLUS PACLITAXEL-CARBOPLATIN VERSUS BEVACIZUMAB PLUS PACLITAXEL-CARBOPLATIN FOR THE FIRST-LINE TREATMENT OF CHINESE PARTICIPANTS WITH ADVANCED NON-SQUAMOUS NON-SMALL CELL LUNG CANCER
Brief Title: A BRIDGING STUDY OF PF-06439535 (CN) PLUS PACLITAXEL-CARBOPLATIN VERSUS BEVACIZUMAB PLUS PACLITAXEL-CARBOPLATIN IN NSCLC
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated as part of the decision by Pfizer to halt its biosimilars programs in China.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B7391007
Record Dates: First submitted 2019-10-14; First posted 2020-03-27 (Actual); Results first posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-06

CONDITIONS: Advanced Non-squamous NSCLC
MeSH Terms: interventions — Bevacizumab; Paclitaxel; Carboplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): PF-06439535 (CN) + paclitaxel + carboplatin
  Interventions: Drug: PF-06439535 (CN); Drug: Paclitaxel; Drug: Carboplatin
- Arm B (Active Comparator): Bevacizumab-EU + paclitaxel + carboplatin
  Interventions: Drug: Bevacizumab-EU; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: PF-06439535 (CN) — 15 mg/kg, IV on day 1 of each 21 day cycle for up to 2 years, or until progression or unacceptable toxicity develops.
  Arms: Arm A
Drug: Bevacizumab-EU — 15 mg/kg, IV on day 1 of each 21 day cycle until disease progression, unacceptable toxicity or 25 weeks. At Week 25, the participants with clinical benefit will received PF-06439535 (CN) monotherapy for up to 2 years from randomization in this study
  Other Names: Avastin
  Arms: Arm B
Drug: Paclitaxel — 175 mg/m2 via IV infusions on Day 1 of a 21-day cycle for each of at least 4 and no more than six (6) 21-day cycles.
Drug: Carboplatin — AUC 5 (max=750mg) via IV infusions on Day 1 of a 21-day cycle for each of at least 4 and no more than six (6) 21-day cycles.

SUMMARY:
The current study will compare the efficacy, safety, pharmacokinetics and immunogenicity of PF-06439535 (CN) in combination with paclitaxel and carboplatin versus bevacizumab sourced from the European Union (bevacizumab-EU) with paclitaxel and carboplatin in Chinese participants with advanced non-squamous NSCLC in the first-line treatment setting.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants age at least 18 years of age.
* Newly diagnosed Stage IIIB, IIIC or IV non small cell lung cancer (NSCLC) (according to American Joint Committee on Cancer (AJCC) Staging Manual, 8th Edition, last updated 05 June 2018) or recurrent NSCLC.
* Histologically or cytologically confirmed diagnosis of non-squamous NSCLC.
* At least one measurable lesion as defined by RECIST v1.1.
* Be eligible to receive bevacizumab, paclitaxel, and carboplatin based on local standard of care, for the treatment of advanced or metastatic non-squamous NSCLC.

Exclusion Criteria:

* Small cell lung cancer (SCLC) or combination SCLC and NSCLC. Squamous-cell tumors and mixed adenosquamous carcinomas.
* Evidence of a tumor that compresses or invades major blood vessels or tumor cavitation that, in the opinion of the investigator, is likely to bleed.
* Known EGFR activating mutations (for example, exon 19 deletion or exon 21 L858R substitution mutations) or ALK rearrangements.
* Prior systemic therapy for advanced NSCLC; prior neoadjuvant or adjuvant therapy is allowed if surgical resection for primary disease was performed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-06-11 (Actual); Primary Completion 2021-05-10 (Actual); Study Completion 2021-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- China (4):
  - Dongguan People's Hospital, Dongguan, Guangdong
  - Affiliated Hospital of Hebei University, Baoding, Hebei
  - Jinan Central Hospital, Jinan, Shandong
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7391007

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was terminated on 17 March 2021 by the Sponsor. This study was conducted in China.
Pre-assignment Details: A total of 13 participants were screened, of which 5 were screen failure. Four participants were randomized into each of the PF-06439535 (CN) or bevacizumab (EU) groups. Sample size after termination is very small. To avoid the risk of participant re-identification, participant flow was reported in a single overall study period.
Groups:
- PF-06439535 (CN): Participants received PF-06439535 (CN) (starting dose of 15 mg/kg) plus paclitaxel (starting dose of 175 mg/m^2) and carboplatin (starting dose of area under the concentration versus time curve [AUC] 5 [max=750 mg]) for up to but not including 25 weeks, followed by PF-06439535 (CN) monotherapy up to 2 years from randomization. Paclitaxel, carboplatin and PF-06439535 (CN) were administered via intravenous (IV) infusion in order on 21-day cycles.
- Bevacizumab (EU): Participants received bevacizumab (EU) (starting dose of 15 mg/kg) plus paclitaxel (starting dose of 175 mg/m^2) and carboplatin (starting dose of AUC 5 [max=750 mg]) for up to but not including 25 weeks, followed by PF-06439535 (CN) monotherapy up to 2 years from randomization. Paclitaxel, carboplatin and bevacizumab (EU) were administered via IV infusion in order on 21 day cycles.
Period: Overall Study
Arm/Group | PF-06439535 (CN) | Bevacizumab (EU)
Started | 4 | 4
Completed | 3 | 1
Not Completed | 1 | 3
Not completed — Study Terminated By Sponsor | 1 | 1
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- PF-06439535 (CN): Participants received PF-06439535 (CN) (starting dose of 15 mg/kg) plus paclitaxel (starting dose of 175 mg/m^2) and carboplatin (starting dose of AUC 5 [max=750 mg]) for up to but not including 25 weeks, followed by PF-06439535 (CN) monotherapy up to 2 years from randomization. Paclitaxel, carboplatin and PF-06439535 (CN) were administered via IV infusion in order on 21 day cycles.
- Total: Total of all reporting groups
Arm/Group | PF-06439535 (CN) | Bevacizumab (EU) | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Customized [Number; unit: Participants] | NA — Data cannot be reported because doing so would risk re-identification of participants. There were very limited participant numbers in each arm. | NA — Data cannot be reported because doing so would risk re-identification of participants. There were very limited participant numbers in each arm. | NA — Data cannot be reported because doing so would risk re-identification of participants. There were very limited participant numbers in each arm.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | NA — Data cannot be reported because doing so would risk re-identification of participants. There were very limited participant numbers in each arm. | NA — Data cannot be reported because doing so would risk re-identification of participants. There were very limited participant numbers in each arm. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Male | NA — Data cannot be reported because doing so would risk re-identification of participants. There were very limited participant numbers in each arm. | NA — Data cannot be reported because doing so would risk re-identification of participants. There were very limited participant numbers in each arm. | NA — Total not calculated because data are not available (NA) in one or more arms.
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 4 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Objective Response
Description: Objective response referred to complete response (CR) or partial response (PR) by Week 19 of the study in accordance with Response Evaluation Criteria in Solid Tumors (RECIST) v 1.1 which was subsequently confirmed by Week 25. A participant achieved CR if both target and non-target lesions achieved CR, no new lesions; achieved PR if target lesions achieved CR or PR, non-target lesions were assessed as non-CR/non-PD (non-progressive disease), indeterminate or missing, and no new lesions. For target lesions, CR: complete disappearance of all target lesions, normal nodes (target nodes must decrease to normal size); PR: >= 30% decrease under baseline of the sum of diameters of all target measurable lesions. For non-target lesions, CR: disappearance of all non-target lesions and normalization of tumor marker levels and all lymph nodes must be normal in size; non-CR/non-PD: persistence of any non-target lesions and/or tumor marker level above the normal limits.
Time Frame: From Week 1 to Week 25 (25 Weeks)
Population: The Intent-to-treat (ITT) population was defined as all participants who were randomized to study treatment. Data for analyzing endpoint were not collected.
Groups:
- PF-06439535 (CN): Participants received PF-06439535 (CN) (starting dose of 15 mg/kg) plus paclitaxel (starting dose of 175 mg/m^2) and carboplatin (starting dose of AUC 5 [max=750 mg]) for up to but not including 25 weeks as treatment period, followed by PF-06439535 (CN) monotherapy up to 2 years from randomization as extension period. Paclitaxel, carboplatin and PF-06439535 (CN) were administered via IV infusion in order on 21 day cycles.
- Bevacizumab (EU): Participants received bevacizumab (EU) (starting dose of 15 mg/kg) plus paclitaxel (starting dose of 175 mg/m^2) and carboplatin (starting dose of AUC 5 [max=750 mg]) for up to but not including 25 weeks as treatment period, followed by PF-06439535 (CN) monotherapy up to 2 years from randomization as extension period. Paclitaxel, carboplatin and bevacizumab (EU) were administered via IV infusion in order on 21 day cycles.
Arm/Group | PF-06439535 (CN) | Bevacizumab (EU)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) in Treatment Period
Description: TEAE was defined as any adverse event that occurs after the beginning of the investigational product or any pre-existing adverse event (AE) that worsens after the beginning of the investigational product. Serious adverse events (SAE) were assessed by the investigator. Severity of AE was graded based on National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03: Grade 3-SEVERE AE; Grade 4-LIFE-THREATENING consequences; urgent intervention indicated; Grade 5-DEATH RELATED TO AE.
Time Frame: From Day 1 to end of Cycle 8; 1 Cycle = 21 Days
Population: The safety population was defined as all participants who were randomized and received at least one dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06439535 (CN) | Bevacizumab (EU)
Number analyzed (Participants) | 4 | 4
Participants
  Participants with all causalities AEs | 4 | 4
  Participants with all causalities SAEs | 1 | 2
  Participants with all causalities AEs of maximum grade 3 or 4 | 2 | 3
  Participants with all causalities AEs of maximum grade 5 | 0 | 0
  Participants with PF-06439535 (CN) or bevacizumab (EU)-related AEs | 4 | 4
  Participants with PF-06439535 (CN) or bevacizumab (EU)-related SAEs | 0 | 1
  Participants with PF-06439535 (CN) or bevacizumab (EU)-related AEs of maximum grade 3 or 4 | 1 | 2
  Participants with PF-06439535 (CN) or bevacizumab (EU)-related AEs of maximum grade 5 | 0 | 0

3. Secondary Outcome: Number of Participants With Anti-Drug Antibodies (ADA)
Description: ADA have been evaluated in studies with bevacizumab in cancer patient populations. A sensitive and specific immunoassay for detecting ADA in human serum was used to analyze the ADA samples (blood samples for assessment of ADA collected at specified timepoints).
Time Frame: Pre-dose on Day 1 of Cycle 1 and Cycle 5, and before the last administration of the investigational product (up to Cycle 14 Day 1); 1 Cycle = 21 Days
Population: All participants who were randomized and received at least 1 dose of investigational product were used for ADA and neutralizing antibody (NAb) analyses. The number of participants analyzed are those numbers with participants ADA samples tested.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06439535 (CN) | Bevacizumab (EU)
Number analyzed (Participants) | 4 | 4
Participants
  Cycle 1_Day 1_ADA Positive | 0 | 0
  Cycle 5_Day 1_ADA Positive: number analyzed (Participants) | 3 | 4
  Cycle 5_Day 1_ADA Positive | 0 | 0
  End of Treatment Positive: number analyzed (Participants) | 4 | 2
  End of Treatment Positive | 0 | 0

4. Secondary Outcome: Number of Participants With NAb
Description: Blood samples for assessment of ADA and NAb were collected at specified time point. Samples that were determined positive for ADA were further characterized for NAb using a single validated NAb assay.
Time Frame: as for outcome 3
Population: All participants who were randomized and received at least one dose of investigational product were used for ADA and NAb analyses. NAb were not tested thus no data were reported. Only samples that were determined positive for ADA would be further characterized for NAb.
Arm/Group | PF-06439535 (CN) | Bevacizumab (EU)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Trough and Apparent Peak PF-06439535 (CN) and Bevacizumab (EU) Concentrations
Description: The drug concentrations were determined using serum samples collected at the time points specified.
Time Frame: Pre-dose on Day 1 of Cycle 1 and Cycle 5, and before the last administration of the investigational product (up to Cycle 14 Day 1); 2.5 hours after initiation of bevacizumab infusion on Day 1 of Cycle 1 and Cycle 5; 1 Cycle = 21 Days
Population: Participants who were randomized and had at least 1 post dose drug concentration measurement, and had no major protocol deviations which influenced the pharmacokinetic (PK) assessment were included in the PK analysis. Data for analyzing endpoint were not collected.
Arm/Group | PF-06439535 (CN) | Bevacizumab (EU)
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Number of Participants With TEAEs in Extension Period
Description: Treatment emergent adverse event (TEAE) was defined as any adverse event that occurs after the beginning of the investigational product or any pre-existing adverse event that worsens after the beginning of the investigational product. Serious adverse events were assessed by the investigator. Severity of AE was graded based on NCI CTCAE version 4.03: Grade 3-SEVERE AE; Grade 4-LIFE-THREATENING consequences; urgent intervention indicated; Grade 5-DEATH RELATED TO AE.
Time Frame: Cycle 9 Day 1 up to End of Treatment (up to Cycle 14 Day 21); 1 Cycle = 21 Days
Population: The safety population was defined as all participants who were randomized and received at least one dose of investigational product. To avoid risk re-identification of participants, data for extension period were reported in 1 arm as a total.
Measure: Count of Participants; unit: Participants
Groups:
- Extension Period: PF-06439535 (CN) or Bevacizumab (EU) > PF-06439535 (CN): Participants in extension period who received PF-06439535 (CN) or bevacizumab (EU) (starting dose of 15 mg/kg) plus paclitaxel (starting dose of 175 mg/m*2) and carboplatin (starting dose of AUC 5 [max=750mg]) for up to but not including 25 weeks as treatment period, followed by PF-06439535 (CN) monotherapy up to 2 years from randomization as extension period. Paclitaxel, carboplatin and PF-06439535 (CN) were administered via IV infusion in order on 21-day cycles.
Arm/Group | Extension Period: PF-06439535 (CN) or Bevacizumab (EU) > PF-06439535 (CN)
Number analyzed (Participants) | 3
Participants
  Participants with all causality AEs | 3
  Participants with all causality SAEs | 1
  Participants with all causality AEs of maximum grade 3 or 4 | 1
  Participants with all causality AEs of maximum grade 5 | 0
  Participants with PF-06439535 (CN) or bevacizumab (EU)-related AEs | 2
  Participants with PF-06439535 (CN) or bevacizumab (EU)-related SAEs | 0
  Participants with PF-06439535 (CN) or bevacizumab (EU)-related AEs of maximum grade 3 or 4 | 1
  Participants with PF-06439535 (CN) or bevacizumab (EU)-related AEs of maximum grade 5 | 0

ADVERSE EVENTS:
Time Frame: From ICD through and up to 28 days after last dose of investigational product or prior to the start of new anticancer therapy, whichever occurred first (up to 311 days).
Description: To avoid risk re-identification of participants, data for extension period were reported in 1 arm as a total.
Groups:
- Treatment Period: PF-06439535 (CN): Participants received PF-06439535 (CN) (starting dose of 15 mg/kg) plus paclitaxel (starting dose of 175 mg/m^2) and carboplatin (starting dose of AUC 5 [max=750 mg]) for up to but not including 25 weeks as treatment period, followed by PF-06439535 (CN) monotherapy up to 2 years from randomization as extension period. Paclitaxel, carboplatin and PF-06439535 (CN) were administered via IV infusion in order on 21-day cycles.
- Treatment Period: Bevacizumab (EU): Participants received bevacizumab (EU) (starting dose of 15 mg/kg) plus paclitaxel (starting dose of 175 mg/m^2) and carboplatin (starting dose of AUC 5 [max=750 mg]) for up to but not including 25 weeks as treatment period, followed by PF-06439535 (CN) monotherapy up to 2 years from randomization as extension period. Paclitaxel, carboplatin and bevacizumab (EU) were administered via IV infusion in order on 21-day cycles.
Arm/Group | Treatment Period: PF-06439535 (CN) | Treatment Period: Bevacizumab (EU) | Extension Period: PF-06439535 (CN) or Bevacizumab (EU) > PF-06439535 (CN)
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 1/4 | 2/4 | 1/3
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Period: PF-06439535 (CN) (N=4) | Treatment Period: Bevacizumab (EU) (N=4) | Extension Period: PF-06439535 (CN) or Bevacizumab (EU) > PF-06439535 (CN) (N=3)
Neutropenia (Blood and lymphatic system disorders) | 1 | 2 | 0
Pyrexia (General disorders) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Period: PF-06439535 (CN) (N=4) | Treatment Period: Bevacizumab (EU) (N=4) | Extension Period: PF-06439535 (CN) or Bevacizumab (EU) > PF-06439535 (CN) (N=3)
Anaemia (Blood and lymphatic system disorders) | 3 | 1 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 0
Nausea (Gastrointestinal disorders) | 2 | 2 | 1
Toothache (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0
Malaise (General disorders) | 1 | 1 | 0
Pain (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 1 | 1
Temperature intolerance (General disorders) | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 1 | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 3 | 1
Platelet count decreased (Investigations) | 2 | 1 | 0
Weight increased (Investigations) | 1 | 1 | 0
White blood cell count decreased (Investigations) | 3 | 3 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 2 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 2 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 0 | 2
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Anaesthesia (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 1 | 0
Neurotoxicity (Nervous system disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0
Merycism (Psychiatric disorders) | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 1 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 3 | 0
Hypertension (Vascular disorders) | 2 | 2 | 1
Fatigue (General disorders) | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
The study was terminated on 17 March 2021 by the Sponsor. The decision to terminate this study was based on a business review of the biosimilars market and the Sponsor's global manufacturing network. This decision was not based on any safety or regulatory concerns with the treatment of participants with PF-06439535 (CN). The results reported are limited to safety, PK and immunogenicity, and only safety is summarized.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2019-06-27): https://cdn.clinicaltrials.gov/large-docs/98/NCT04325698/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-05): https://cdn.clinicaltrials.gov/large-docs/98/NCT04325698/SAP_001.pdf